CLINICAL TRIAL: NCT04654117
Title: Examining the Active Ingredients of Consultation to Improve Implementation of a Parent-mediated Intervention for Children With Autism in the Community Mental Health System
Brief Title: Examining the Active Ingredients of Consultation of a Parent-mediated Intervention for Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Brooke Ingersoll, Professor of Psychology, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R40MC27705
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Consultation; Autism Spectrum Disorder; Medicaid; Parent-mediated intervention; Parent Training
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): Following completing the online tutorial, each agency will have a baseline lasting 3-6 weeks (this will be staggered by agency).
- Treatment (Consultation) (Experimental): Consultation will be conducted in 4-week phases that correspond to the three consultation components. The phases will occur in a randomized order. During a given phase, no components of any other phases will be provided. Feedback phase. Consultees will submit 5-minute clips of session recordings of their Project ImPACT session with their enrolled family for feedback. Oral feedback will be provided by the consultant and peers. Case support phase. The consultant will lead the group in problem-solving common barriers that providers experience with their cases. Skill rehearsal phase. The consultant will lead skill rehearsal practices in which providers role play elements of a Project ImPACT session.
  Interventions: Other: Consultee-centered administrative consultation
- Follow Up (No Intervention): During the follow-up period, consultation will not occur, and providers will continue implementing Project ImPACT with their cases. Eight weeks post-consultation, providers will submit a recorded Project ImPACT session with their enrolled family. Providers and caregivers will complete a final online questionnaire.

INTERVENTIONS:
Other: Consultee-centered administrative consultation — The consultee-centered administrative consultation model expressly focuses on supporting providers to increase EBP implementation within their specific setting.
  Arms: Treatment (Consultation)

SUMMARY:
Parent-mediated interventions are considered best practice for treating children with autism spectrum disorder, but these interventions are underutilized in community settings. Implementation strategies like consultation can improve the implementation of these interventions, but little is known about the active ingredients of consultation. This study uses an experimental design (ABCD single-case design with multiple baselines) to identify the active ingredients of a consultation model designed to support the implementation of a parent-mediated intervention for autism spectrum disorder in a low-resourced community mental health system.

DETAILED DESCRIPTION:
There are multiple evidence-based practices (EBPs) to treat autism spectrum disorder (ASD), yet the gap from when EBPs are developed to when they reach community settings is 17 years. EBPs are consistently underused in community settings despite their well-studied effectiveness. One such EBP for treating ASD in young children is parent-mediated intervention.

Consultation is one method of supporting implementation that involves providing clinicians with support and feedback from intervention experts. For this study, consultation on an evidence-based parent-mediated intervention, Project ImPACT, will be the focus. Understanding the active ingredients that go into consultation is important to understand how consultation works so that it can be tailored to best meet the needs of community settings. This single-case experimental design (SCED) will manipulate three potential ingredients of consultation: feedback on taped sessions, case support, and skill rehearsal.

Groups of 3-5 providers per agency will be given 2 weeks to complete a 6-hour self-directed online tutorial on Project ImPACT utilized regularly by Project ImPACT consultants. Next, each agency will be randomly assigned to baselines lasting 3-6 weeks, followed by 4 weeks of each consultation component (total of 12 weeks). All agencies will receive consultation. The order of the consultation components will be randomized using a random number generator such that each agency has an equal chance of receiving one of the predetermined permutations of phases which are labeled in alphabetical order (e.g., equally as likely to be randomized to ABCD order as ADBC order). Across each phase, providers will record one session per week with their enrolled family and submit it via a HIPAA-compliant Drop-box link. Providers will complete weekly online questionnaires on implementation outcomes, with time reserved during consultation sessions to complete them. After consultation, providers will submit a final recorded session and questionnaire 8-weeks post-consultation. Caregivers will complete a measure of social communication for their child via online questionnaire at baseline, twice during consultation, and after 8 weeks post-consultation.

The feedback phase will involve the consultant and peers responding to the 5-minute clips of recorded telehealth sessions with praise and constructive feedback. The case support phase will be a time for the consultant and peers to assist in any challenges faced; for example, this could include issues with telehealth, caregiver coaching, or family/child needs. The skill rehearsal phase will allow for consultees to practice their clinical skills via role play.

This study will have 4 aims:

Specific Aim 1: Identify the potential active ingredients of the consultation model by evaluating its effects on providers' treatment adherence and parent-mediated intervention competence. The investigators predict that the feedback component will improve adherence and competence over and above improvements from the case support and skill rehearsal components.

Specific Aim 2: Examine the relative feasibility, acceptability, and appropriateness of each consultation component using a SCED component analysis. Feasibility is the extent to which a practice can be successfully carried out within a setting. Acceptability is the extent to which a practice is agreeable and satisfactory. Appropriateness is the perceived fit or relevance of a practice to address a problem. The investigators predict that providers will perceive the case support component to be the most feasible, acceptable, and appropriate of all components.

Specific Aim 3: Examine the effects of the consultation model on case penetration and the feasibility, acceptability, and appropriateness of the EBP (Project ImPACT). The investigators predict case penetration (i.e., total number of Project ImPACT cases on a provider's caseload divided by the total number of eligible clients) and EBP feasibility, acceptability, and appropriateness to increase over time.

Exploratory Aim 4: Demonstrate associated social communication outcomes for Medicaid-enrolled children with ASD from baseline to post-consultation. Given that consultation leads to improved adherence and child outcomes and Project ImPACT results in improved child social communication outcomes, the investigators predict that our consultation model will be associated with improvements in child social communication skills.

ELIGIBILITY:
Groups of 3-5 providers will be recruited from four applied behavior analysis (ABA) agencies (~20 providers in total) that contract with regional community mental health agencies to provide ABA services to Medicaid-enrolled children with autism spectrum disorder (ASD). Families on the providers' caseloads will be enrolled.

Inclusion Criteria for Providers:

• Have at least one caregiver on their caseload who would be appropriate for Project ImPACT and who agrees to enroll in the study and have their sessions recorded.

Exclusion Criteria for Providers:

* Not qualified to bill for ABA services through the Medicaid Autism Benefit.
* Under age 18

Inclusion Criteria for Caregivers:

* Parent or guardian of a child who has a community diagnosis of ASD established using the Autism Diagnostic Observation Schedule (a gold standard ASD assessment), receives services through the Medicaid Autism Benefit (requires a household income at or below 133% of the federal poverty line), is between the ages of 18 months and 6 years, which is the age range targeted for Project ImPACT, and has at least 1 session per week with the provider.
* Child's provider is enrolled in the study.

Exclusion Criteria for Caregivers:

• Under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Ingersoll, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Provider Treatment (Consultation): All providers received consultation. Consultation was conducted in 4-week phases that correspond to the three consultation components: Case Support, Feedback, and Skill Rehearsal. The phases will occur in a randomized order. During a given phase, no components of any other phases were provided. Feedback phase. Consultees submitted 5-minute clips of session recordings of their Project ImPACT session with their enrolled family for feedback. Oral feedback was provided by the consultant and peers. Case support phase. The consultant led the group in problem-solving common barriers that providers experience with their cases. Skill rehearsal phase. The consultant led skill rehearsal practices in which providers role played elements of a Project ImPACT session.
- Family Treatment (Project ImPACT): All families received Project ImPACT. Project ImPACT is an evidence-based manualized parent coaching program that is designed to teach caregivers strategies to support social communication development in young children with autism or social communication delays. Project ImPACT is a naturalistic developmental behavioral intervention (NDBI), which is a newer class of autism intervention that blends principles of developmental science and applied behavior analysis (Schreibman et al., 2015). Clinicians were instructed to deliver the Project ImPACT program once per week via a telehealth platform supported by their agency (e.g., Zoom, HIPAA-compliant Google Meet), for a total of 24 sessions, with a session length of 60 minutes per session.
Period: Overall Study
Arm/Group | Provider Treatment (Consultation) | Family Treatment (Project ImPACT)
Started | 20 | 21
Completed | 16 | 13
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Provider Treatment (Consultation) | Family Treatment (Project ImPACT) | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Full Range); unit: years] | 32 [23 to 58] | 36 [23 to 54] | 35 [23 to 58]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 caregivers had missing data for sex.
  Participants
    number analyzed (Participants) | 20 | 19 | 39
    Female | 18 | 17 | 35
    Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 caregivers had missing data for ethnicity.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 20 | 19 | 39
    Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 caregivers had missing data for race.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 4 | 4
    White | 20 | 14 | 34
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 2 | 2
Project ImPACT Coaching Fidelity [Mean (Full Range); unit: units on a scale] — The Project ImPACT Coaching Fidelity Checklist is a measure of treatment adherence. It uses a 3-point scale -- Observed (1), Partially Observed (.5), and Not Observed (0). Higher scores indicate higher treatment adherence. Based on scoring guidelines for this measure, scores for each item are multiplied by an item-specific weight value. Scores for each item are then summed and divided by the total number of items scored, yielding a score ranging from 0 to 100. Population: This measure is only for providers and refers to their fidelity to using Project ImPACT.
  units on a scale
    number analyzed (Participants) | 20 | 0 | 20
    (all) | 62.51 [25 to 94] |  | 62.51 [25 to 94]
PEACE Parent Coaching Competency Fidelity [Mean (Full Range); unit: units on a scale] — Parent-mediated intervention competence will be assessed via Parent Empowerment and Coaching in Early Intervention (PEACE) coding which utilizes a 5-point scale to assess for competency in delivering collaborative coaching techniques used in parent-mediated interventions. The scale used is: Never (1), Rarely (2), Sometimes (3), Often (4), and Almost Always (5). The minimum value on the scale is 1 and the maximum is 5. Higher scores indicate higher parent-mediated intervention competence. Population: This measure is only completed for providers, as it is a measure of competency in delivering parent coaching interventions.
  units on a scale
    number analyzed (Participants) | 20 | 0 | 20
    (all) | 2.87 [1.53 to 4.24] |  | 2.87 [1.53 to 4.24]
Autism Impact Measure [Mean (Full Range); unit: units on a scale] — The Autism Impact Measure has 41 items rated based on the sum of scores on two scales (frequency and impact) that both include a 5-point scale ranging from Never (1) to Always (5). Higher values indicate higher frequency of concerns and higher impact of concerns on child functioning. The minimum value is 82 and the maximum value is 410. Population: This measure was only for caregivers as it is a caregiver-report questionnaire of child skills.
  units on a scale
    number analyzed (Participants) | 0 | 21 | 21
    (all) |  | 234.76 [122 to 313] | 234.76 [122 to 313]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence
Description: The Project ImPACT Coaching Fidelity Checklist is a measure of treatment adherence. It uses a 3-point scale -- Observed (1), Partially Observed (.5), and Not Observed (0). Higher scores indicate higher treatment adherence. Based on scoring guidelines for this measure, scores for each item are multiplied by an item-specific weight value. Scores for each item are then summed and divided by the total number of items scored, yielding a score ranging from 0 to 100.
Time Frame: 23-26 weeks
Population: This measure is only collected from the provider arm.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Providers: Al providers in the study submitted telehealth sessions and a series of questionnaires.
Arm/Group | Providers
Number analyzed (Participants) | 12
score on a scale | 62.51 (5.08)
Statistical Analysis 1: Comparison: Providers; Test type: Superiority — Multilevel model predicting the effect of the overall consultation model on manual adherence, averaged across clinicians; p < .05, multilevel model; unstandardized beta = 0.33, Standard Error of Mean 3.85

2. Primary Outcome: Parent-mediated Intervention Competence
Description: Parent-mediated intervention competence will be assessed via Parent Empowerment and Coaching in Early Intervention (PEACE) coding which utilizes a 5-point scale to assess for competency in delivering collaborative coaching techniques used in parent-mediated interventions. The scale used is: Never (1), Rarely (2), Sometimes (3), Often (4), and Almost Always (5). The minimum value on the scale is 1 and the maximum is 5. Higher scores indicate higher parent-mediated intervention competence.
Time Frame: 23-26 weeks
Population: This measure is only collected from the provider arm.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Providers
Number analyzed (Participants) | 12
score on a scale | 2.87 (0.11)
Statistical Analysis 1: Comparison: Providers; Test type: Superiority; p < .05, multilevel model; unstandardized beta = 0.04, Standard Error of Mean 0.08

3. Primary Outcome: Case Penetration
Description: Case penetration will be measured weekly using the Penetrability Formula and will be expressed using provider report of the total number of Project ImPACT cases on their caseload divided by the total number of eligible clients with ASD on their Medicaid Autism Benefit caseload. This is expressed as a percentage. Higher percentage values indicate higher case penetration.
Time Frame: 23-26 weeks
Population: This measure is only collected from the provider arm. 288 observations (i.e., surveys) across 20 clinicians from 6 agencies were included in the models.
Measure: Mean (Standard Error); unit: percentage of caseload
Groups:
- Providers: Al providers in the study submitted telehealth sessions and a series of questionnaires. Case penetration for clients using Medicaid insurance was measured using the Penetrability Formula.
Arm/Group | Providers
Number analyzed (Participants) | 20
percentage of caseload | 24.37 (4.48)
Statistical Analysis 1: Comparison: Providers; Test type: Other — multilevel modeling; p < .05, multilevel modeling; multilevel modeling = 2.56, Standard Error of Mean 0.74

4. Primary Outcome: Ratings of the Usability of Each Consultation Component
Description: Clinicians reported on the usability of each consultation component weekly across the 4 weeks of each consultation condition using the Implementation Strategy Usability Scale (Lyon et al., 2021). This 10-item questionnaire uses a 5-point Likert scale to examine clinician perceptions about the complexity of using an implementation strategy. The scale is unidimensional and has no subscales. Based on scoring guidelines, a formula is used to calculate the total usability score, which ranges from 0-100. Higher scores indicate higher usability; higher scores indicate higher ratings of the participant's ability to use the strategy with ease. The formula involves the following: for each odd numbered item, subtract 1 from the Likert rating value to get the new value; for each even numbered item, subtract the Likert rating value from 5 to get a new value; then sum all new values and multiply by 2.5.
Time Frame: 23-26 weeks
Population: This measure is only collected from the provider arm. 20 clinicians reported on usability of each consultation component.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Providers: All providers in the study submitted telehealth sessions and a series of questionnaires.
Arm/Group | Providers
Number analyzed (Participants) | 20
score on a scale
  Case Support | 76.78 (14.12)
  Skill Rehearsal | 60.71 (15.99)
  Feedback on Videotaped Sessions | 72.01 (15.37)
Statistical Analysis 1: Comparison: Providers; Test type: Superiority; p < .05, ANOVA; ANOVA = 17.00

5. Primary Outcome: Ratings of Perceptions of Project ImPACT
Description: Providers completed the Perceived Characteristics of Intervention Scale (PCIS; Cook et al., 2015) weekly about their perceptions of Project ImPACT. This 18-item questionnaire includes items related to various constructs from Rogers' Diffusions of Innovation theory (Rogers, 2010). All items are rated on a 7-point Likert scale and the overall PCIS score is established by computing the mean of all items. The minimum score is 1.00 and maximum is 7.00. Higher values indicate more positive perceptions of the intervention.
Time Frame: 23-26 weeks
Population: This measure is only collected from the provider arm. 286 surveys from 18 clinicians with sufficient data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Providers
Number analyzed (Participants) | 18
score on a scale | 3.38 (0.18)
Statistical Analysis 1: Comparison: Providers; Test type: Other — multilevel model; p < .05, multilevel model; multilevel model = 0.04, Standard Error of Mean 0.02

6. Primary Outcome: Child Social Communication Skills
Description: The Autism Impact Measure has 41 items rated on a 5-point scale ranging from Never (1) to Always (5). The overall score is calculated by summing the scores on two scales (frequency and impact). Higher values indicate a higher frequency and impact of autism-related concerns child functioning. The minimum value is 82 and the maximum value is 410.
Time Frame: 23-26 weeks
Population: This measure is only collected from the caregiver arm (caregivers reporting on child skills). Models included 62 surveys across 17 children from 5 agencies.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Families: Caregivers reported on child skills throughout the intervention period.
Arm/Group | Families
Number analyzed (Participants) | 17
score on a scale | 40.09 (2.70)
Statistical Analysis 1: Comparison: Families; Test type: Other — multilevel model; p < .05, multilevel model; multilevel model (beta) = -0.27, Standard Error of Mean 0.15

ADVERSE EVENTS:
Time Frame: 23-27 weeks
Description: This was an observational study of a psychosocial intervention provided in routine behavioral health settings. No adverse events occurred during the course of the study.
Arm/Group | Provider Treatment (Consultation) | Family Treatment (Project ImPACT)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT04654117/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT04654117/ICF_000.pdf